CLINICAL TRIAL: NCT00810654
Title: Study on The Effectiveness of Oral Administration of Prolyl Endoprotease for Gluten Detoxification as a Means to Treat Coeliac Disease
Brief Title: Effect of Aspergillus Niger Prolyl Endoprotease (AN-PEP) Enzyme on the Effects of Gluten Ingestion in Patients With Coeliac Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: DSM Food Specialties (Industry); Leiden University Medical Center (Other)
Responsible Party: C.J.Mulder, VU University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RD.0601.54; NTR1281
Record Dates: First submitted 2008-12-17; First posted 2008-12-18 (Estimated); Last update posted 2011-01-19 (Estimated); Status verified 2009-05

CONDITIONS: Celiac Disease
Keywords: Celiac disease; Coeliac disease; treatment; AN-PEP; prolyl endoprotease; gluten
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ANPEP (Experimental): Aspergillus niger prolyl endoprotease (AN-PEP), a microbial-derived prolyl endoprotease which cleaves gluten
  Interventions: Dietary Supplement: Aspergillus niger prolyl endoprotease
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Aspergillus niger prolyl endoprotease — 160 PPU daily for 2 weeks
  Other Names: AN-PEP
  Arms: ANPEP
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Oral supplementation with enzymes that can cut gluten has been suggested as a potential treatment modality for coeliac disease. In the present study the investigators wish to determine if co-administration of such an enzyme, a prolyl endoprotease derived from the food grade organism Aspergillis niger (AN-PEP), is capable of detoxifying 8 grams of gluten in a commercial food product.

DETAILED DESCRIPTION:
The objective of the study is to determine whether AN-PEP enzyme is effective in mitigating the effects of 8 g wheat protein ingestion in patients with celiac disease.

Fourteen patients with coeliac disease, 18-70 years old are recruited. During the first period, patients consume once daily a gluten-containing food product with the AN-PEP enzyme for 2 weeks. After a 2-week washout period (second period), patients enter the third period of this study, and are randomized to one of two groups and consume the same gluten-containing food product with AN-PEP or placebo.

Period 1: Patients are given a food product containing 8 g of wheat protein, to which AN-PEP is added, once daily for 14 d.

Period 2: Wash-out period of 14 d. During this period, patients will consume a gluten-free diet.

Period 3: Patients who are negative for coeliac disease symptoms during the 1st period will be randomized across two groups. Both groups receive a food product containing 8 g of wheat protein once daily for 14 d. One group receives additional AN-PEP with the gluten meal whereas the other group receives the placebo.

Patients will visit the outpatient clinic five times; one visit before the start of the study, a visit during and at the end of the first period, and a visit during and at the end of the third period. During three of the visits, spike-biopsies are taken from the duodenum by oesophago-gastro-duodenoscopy. Blood samples are taken during all of the five visits. Patients will also fill in a quality of life questionnaire at the start and the end of the first and third period.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of coeliac disease (Marsh III B/C) ; that means crypt hyperplasia and subtotal or total villous atrophy, while using a normal diet followed by normalisation and clinical improvement on a gluten-free diet;
* Detectable coeliac disease specific antibodies (EMA, tTGA) at time of diagnosis.
* A strict gluten free diet for at least 1 year and normalised villous architecture (Marsh 0/I);
* Male and female, 18-70 years old;
* No detectable anti-endomysium and low anti-tissue transglutaminase (< 4 U/ml) prior to the start of the study;
* Patient is willing to undergo all protocol related assessments and visits (including up to 3 separate oesophago-gastro-duodenoscopies with multiple biopsies taken each time from the descending duodenum);
* Patient has read the information provided on the study and given written consent;
* Female participants at fertile age must use adequate contraception.

Exclusion Criteria:

* Use of any immunoregulatory drug within the last 6 months;
* Use of any anticoagulant drug;
* Clinically suspected bleeding tendency;
* Pregnancy or breast feeding;
* Presence of any concurrent active infection;
* IgA deficiency.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2008-05; Primary Completion 2009-05 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Histopathological changes according to the Modified Marsh criteria | One week before start, and 2 and 6 weeks after start
The presence of coeliac disease specific antibodies (EMA, tTGA, gliadin) | One week before start, and 2 and 6 weeks after start

SECONDARY OUTCOMES:
Presence and activity of gluten reactive Tcells isolated from biopsies and serum | One week before start, and 2 and 6 weeks after start
Immunophenotype of lymphocytes isolated from biopsies | One week before start, and 2 and 6 weeks after start
Clinical symptoms after gluten intake with and without AN-PEP | One week before start, and 2 and 6 weeks after start

CONTACTS AND LOCATIONS:
Overall Officials: Greetje J Tack, MD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- VU University Medical Center, Amsterdam, Netherlands

REFERENCES:
- [Derived] Tack GJ, van de Water JM, Bruins MJ, Kooy-Winkelaar EM, van Bergen J, Bonnet P, Vreugdenhil AC, Korponay-Szabo I, Edens L, von Blomberg BM, Schreurs MW, Mulder CJ, Koning F. Consumption of gluten with gluten-degrading enzyme by celiac patients: a pilot-study. World J Gastroenterol. 2013 Sep 21;19(35):5837-47. doi: 10.3748/wjg.v19.i35.5837. PMID 24124328